CLINICAL TRIAL: NCT07158697
Title: Health Chat for Empowerment-based Lifestyle Planning for Cardiometabolic Multimorbidity (HcELP_CMM) Program: a Randomized Controlled Trial Study
Brief Title: Health Chat for Empowerment-based Lifestyle Planning for Cardiometabolic Multimorbidity
Acronym: HcELP_CMM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jing Xi, PhD, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 25-383
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cardiometabolic Diseases; Multimorbidity
Keywords: Cardiometabolic multimorbidity; Empowerment; Patient-centered; Self-management; Intervention
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention group to receive the HcELP_CMM program intervention or a control group to receive the usual care.
Who Masked: Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HcELP_CMM (Experimental): Participants in the arm will attend a 12-week HcELP_CMM program. This program is a hybrid intervention involving two phases: 1) an initial individualized, face-to-face meeting to collaboratively set goals and develop action plan (week 1); 2) an ongoing, personalized online support delivered by WeChat platform utilizing the official account, chat function, and synchronized online videos to integrate and sustain healthy lifestyle (weekly, week 2-12). Phase 1 covers 4 core steps: 1) assess symptom burden and lifestyle behaviors; 2) generate and analysis symptom burden and lifestyle report; 3) empowerment-based therapeutic person-centered health communication; and 4) behavior commitment. Phase 2 covers two modules: 1) integrate healthy behaviors to long-term lifestyle, and 2) sustain healthy lifestyle behaviors.
  Interventions: Behavioral: HcELP_CMM
- Usual care-maintain daily lifestyle (Placebo Comparator): Participants in the arm will continue with their normal daily lifestyle. WeChat-based follow-up will be performed weekly in the first 4 weeks and bi-weekly in the next 8 weeks. Each follow-up will last for 20 minutes. Follow-up communications will include: (1) general well-being assessments using brief, non-intrusive inquiries (e.g., "How have participants felt overall in the past week/two weeks?"); (2) disease management monitoring through standardized question tracking significant changes in their underlying diseases, intentionally avoiding exploration of intervention-targeted lifestyle behaviors (e.g., "Have participants experienced notable changes in their health status or disease management approach since last contact?"); and (3) addressing disease-related inquiries. For any questions inquired by participants in the control group, general advice will be given for ethical consideration.
  Interventions: Behavioral: Usual care-maintain daily lifestyle

INTERVENTIONS:
Behavioral: HcELP_CMM — The intervention consists of two phases. Phase 1 is an initial individualized, face-to-face meeting to collaboratively set goals and develop action plan (week 1) and Phase 2 is an ongoing, personalized online support delivered by WeChat platform utilizing the official account, chat function, and synchronized online videos to integrate and sustain healthy lifestyle (weekly, week 2-12). Phase 1 covers 4 core steps: 1) assess symptom burden and lifestyle behaviors; 2) generate and analysis symptom burden and lifestyle report; 3) empowerment-based therapeutic person-centered health communication; and 4) behavior commitment. Phase 2 covers two modules: 1) integrate healthy behaviors to long-term lifestyle, and 2) sustain healthy lifestyle behaviors.
  Arms: HcELP_CMM
Behavioral: Usual care-maintain daily lifestyle — Participants in this group will continue with their normal daily lifestyle. WeChat-based follow-up will be performed weekly in the first 4 weeks and bi-weekly in the next 8 weeks. Each follow-up will last for 20 minutes. Follow-up communications will include: (1) general well-being assessments using brief, non-intrusive inquiries (e.g., "How have participants felt overall in the past week/two weeks?"); (2) disease management monitoring through standardized question tracking significant changes in their underlying diseases, intentionally avoiding exploration of intervention-targeted lifestyle behaviors (e.g., "Have participants experienced notable changes in their health status or disease management approach since last contact?"); and (3) addressing disease-related inquiries. For any questions inquired by participants in the control group, general advice will be given for ethical consideration.
  Arms: Usual care-maintain daily lifestyle

SUMMARY:
The goal of this study is to:

1. assess the feasibility of the health chat for empowerment-based lifestyle planning for cardiometabolic multimorbidity (HcELP_CMM);
2. examine the immediate effects of the HcELP_CMM program on lifestyle behaviors, cardiometabolic indicators, symptom burden, health-related quality of life (HRQoL), psychological well-being, and physical function;
3. examine the long-term effects of the HcELP_CMM program on lifestyle behaviors, cardiometabolic indicators, symptom burden, HRQoL, psychological well-being, and physical function in patients with CMM.

The main questions it aims to answer are:

1. If the HcELP_CMM program is feasible?
2. If the HcELP_CMM program has the potential to improve the lifestyle behaviors, cardiometabolic indicators, symptom burden, HRQoL, psychological well-being, and physical function in patients with CMM compared to the usual care group in the short-term？
3. If the HcELP_CMM program has the potential to improve the lifestyle behaviors, cardiometabolic indicators, symptom burden, HRQoL, psychological well-being, and physical function in patients with CMM compared to the usual care group in the long-term？

DETAILED DESCRIPTION:
This study has two parts. Part 1 is a sequential mixed-method pilot study consisted of a single-blind, parallel-group, two-arm randomized controlled trial followed by a qualitative descriptive study. Part 2 is a full single-blind, parallel-group, two-arm randomized controlled trial study. In these two parts, participants with CMM will be randomly assigned to either an intervention group to receive the HcELP_CMM intervention or a control group to receive the usual care in a 1:1 ratio.

For part 1, the intervention group will participate in the 12-week HcELP_CMM project. The intervention consists of two phases. Phase 1: It involves an individualized face-to-face meeting conducted by the researcher in a private meeting room at the community health care centers (CHCCs) within one week after random allocation, lasting about 1 hour. This phase includes four core steps: 1) assessing symptom burden and lifestyle behaviors; 2) generating and analyzing a symptom burden and lifestyle report; 3) engaging in empowerment-based therapeutic person-centered health communication; and 4) making a behavior commitment. Phase 2 will be delivered individually through the WeChat platform using the official account, chat function, and synchronized online video between weeks 2 and 12. It includes two modules:1) integrating healthy behaviors into a long-term lifestyle; and 2) sustaining healthy lifestyle behaviors. In Module 1, participants will implement action plans weekly, and a source hub of empowerment videos will be provided to promote the implementation of action plan. Additionally, participants will self-evaluate lifestyle behaviors, fill out and upload the logbook of self-assessment lifestyle behavior weekly. In Module 2, participants will self-monitor bio-feedback parameters, fill out and upload the logbook of self-monitoring biofeedback parameters weekly. Furthermore, they will receive bi-weekly health counseling through synchronized online videos on the WeChat platform, with each session lasting about 20 minutes. The control group will continue with their normal daily lifestyle. WeChat-based follow-ups will be conducted weekly during the first 4 weeks and biweekly in the subsequent 8 weeks, with each follow-up lasting 20 minutes. Follow-up communications will include: general well-being assessments; disease management monitoring; and addressing disease-related inquiries.Outcome data collection will occur in 1 week after the completion of the intervention through face-to-face interviews at the CHCCs, lasting about 30 minutes. Additionally, some participants in the intervention group will undergo semi-structured interviews via synchronized online video through the WeChat platform in1 week after the intervention concludes, lasting 1 hour. The interview will be audio recorded. Outcome data collection will occur in 1 week after the completion of the intervention through face-to-face interviews at the CHCCs, lasting about 30 minutes.

For part 2, the intervention group will participate in the 12-week HcELP_CMM project. The intervention consists of two phases. Phase 1: It involves an individualized face-to-face meeting conducted by the researcher in a private meeting room at the CHCCs within one week after random allocation, lasting about 1 hour. This phase includes four core steps: 1) assessing symptom burden and lifestyle behaviors; 2) generating and analyzing a symptom burden and lifestyle report; 3) engaging in empowerment-based therapeutic person-centered health communication; and 4) making a behavior commitment. Phase 2 will be delivered individually through the WeChat platform using the official account, chat function, and synchronized online video between weeks 2 and 12. It includes two modules:1) integrating healthy behaviors into a long-term lifestyle; and 2) sustaining healthy lifestyle behaviors. In Module 1, participants will implement action plans weekly, and a source hub of empowerment videos will be provided to promote the implementation of action plan. Additionally, participants will self-evaluate lifestyle behaviors and fill out and upload the logbook of self-assessment lifestyle behavior weekly. In Module 2, participants will self-monitor bio-feedback parameters, fill out and upload the logbook of self-monitoring biofeedback parameters weekly. Furthermore, they will receive bi-weekly health counseling through synchronized online videos on the WeChat platform, with each session lasting about 20 minutes. The control group will continue with their normal daily lifestyle. WeChat-based follow-ups will be conducted weekly during the first 4 weeks and biweekly in the subsequent 8 weeks, with each follow-up lasting 20 minutes. Follow-up communications will include: general well-being assessments; disease management monitoring; and addressing disease-related inquiries. Besides, all participants in the intervention and control groups will undergo a 2-month follow-up after the intervention. During the follow-up period, all participants will maintain their daily lifestyle at home and obtained WeChat-based follow-up bi-weekly. Followup communications include: general well-being assessments; disease management monitoring; and addressing disease related inquiries. Outcome data collection will occur in 1 week after the completion of the intervention and follow-up through face-to-face interviews at the CHCCs, lasting about 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or above；
2. Diagnosed with cardiometabolic multimorbidity (CMM) by doctors, which was defined as co-existing with two or more cardiometabolic diseases, including primary hypertension, primary type 2 diabetes, stroke, and heart diseases (eg. ischemic heart disease, arrhythmia, heart valve diseases, and other heart diseases);
3. Possessed a digital device installed with WeChat, as well as with an internet connection.

Exclusion Criteria:

1. Contraindications to exercise according to American College of Sports Medicine (ACSM), such as severe musculoskeletal disorders, severe cardiovascular diseases, or spinal nerve injury;
2. Diagnosis of psychiatric disease;
3. Has impaired cognitive function as indicated by an Abbreviated Mental Test Score (AMTS) ≤6;
4. Has impaired sensory or communication function which hider them participation in this program, such as hearing loss, vision loss, and unable to speak Mandarin;
5. Unable to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Lifestyle behaviors | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be assessed both in the pilot part and full RCT part. Lifestyle behaviors will be measured by the Health Promoting Lifestyle Profile II (HPLP-II). It encompassed 52 items with six aspects of health promotion behaviors including nutrition, interpersonal support, stress management, exercise, health responsibility, and self-actualization. The HPLP-II uses a four-point scale with 1-4 representing always to never with a total score ranging from 52 to 208 and a higher score indicates better health behavior. It has been translated and validated in China, and the Chinese version has a Cronbach's α coefficient from 0.84 to 0.91.

SECONDARY OUTCOMES:
Eligibility rate | Eligibility rate will be assessed at baseline only in the pilot part.
  Eligibility rate will only be measured in the pilot part，which will be calculated as eligible participants divided by screened participants.
Recruitment rate | Recruitment rate will be assessed at baseline only in the pilot part.
  Recruitment rate will only be measured in the pilot part, which will be calculated as randomized participants divided by eligible participants.
Attendance rate | Attendance rate will be assessed through study completion (an average of 12 weeks) in the pilot part only.
  Attendance rate will only be measured in the pilot part，which will be calculated as sessions attended by the participants divided by planned sessions.
Adherence rate | Adherence rate will be assessed through study completion (an average of 12 weeks) in the pilot part only.
  Adherence rate will only be measured in the pilot part, which will be calculated as participants who completed the program divided by randomized participants.
Attrition rate | Attrition rate will be assessed through study completion (an average of 12 weeks) in the pilot part only.
  Attrition rate will only be measured in the pilot part, which will be calculated as participants dropping out divided by randomized participants.
Participant's engagement experiences, feedback about the study design, and perceived program effects | Participant's engagement experiences, feedback about the study design, and perceived program effects will be measured within one week after the completion of the intervention only in the pilot part.
  Participant's engagement experiences, feedback about the study design, and perceived program effects will only be measured in the pilot part, which will be explored by the individualized semi-structured qualitative interviews with participants in the HcELP_CMM group through synchronized online video interviewing via WeChat platform.
Blood pressure | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be assessed in the pilot part and in the full RCT part. Blood pressure will be taken in the sitting position using an electronic sphygmomanometer. Before measurement, patients will be required to sit still for more than 5 min. The average of three consecutive measurements will be considered the effective blood pressure.
Capillary fasting plasma glucose | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be assessed in the pilot part and in the full RCT part, which will be determined by using a Contour TS blood glucose meter and supporting test strips (BAYER, Germany).
Waist circumference | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be assessed in the pilot part and in the full RCT part，which will be measured with a flexible plastic tape measure at the navel position after the patient exhaled.
Body Mass Index | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be assessed in the pilot part and in the full RCT part，which will be calculated for each patient by dividing their weight in kilograms by the square of their height in meters.
Symptom burden | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be assessed in the pilot part and in the full RCT part. It will be assessed by the Memorial Symptom Assessment Scale (MSAS). MSAS includes 32 commonly occurring symptoms experienced during the preceding week in terms of three dimensions - frequency, severity and distress - for 24 symptoms, and two dimensions - severity and distress -for 8 symptoms. The prevalence of each symptom is answered by yes/no; frequency on a four-point scale(1-4): rarely, occasionally, frequently or almost constantly; severity on a four-point scale(1-4): slight, moderate, severe, or very severe; and distress on a five-point scale(0-4) - not at all, a little bit, somewhat, quite a bit or very much. One item related to sexual was excluded because discussing sex can cause discomfort among Chinese participants. The total symptom burden score per patient is the mean of all symptom burden scores.
Health-related quality of life | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be assessed in the pilot part and in the full RCT part. The 12-item Short Form Health Survey (SF-12) will be used to assess the Health-related quality of life. It is a simplified version of the 36-item Short Form Health Survey (SF-36), but it's almost equivalent to SF-36 and easier to understand and complete. It evaluates 8 dimensions, including general health, physical functioning , role-physical, bodily pain for physical component summary, and vitality, social functioning, role-emotional, and mental health for mental component summary. The total score of physical component summary and mental component summary both ranges from 0 to 100, and a higher score means better physical or mental status. SF-12 has good reliability, content, and construct validity.
Depression | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be assessed in the pilot part and in the full RCT part. Depression will be measured with the Chinese version of the Patient Health Questionnaire-9 (PHQ-9). The scale comprises nine items, with each item rated on a 4-point scale from 0 (not at all) to 3 (almost every day). The total score ranges from 0 to 27, with higher scores indicating more severe depression. The cut-off points of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively. In this study, we used a score of 5 as the cut-off point, with a score greater than or equal to 5 indicating the presence of depressive symptoms. The Cronbach's α coefficient of the total scale is 0.86 for the Chinese general population.
Handgrip | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be measured in the pilot part and in the full RCT part, which will be measured twice by a dynamometer in the dominant hand and the maximum value will be recorded.
5-times-sit-to-stand test | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be measured in the pilot part and in the full RCT part. Participants will be asked to stand up straight and sit as fast as possible on a standard-height chair without armrests, five times without stopping. The completion time will be recorded.
Time up-and-go test | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be measured in the pilot part and in the full RCT part. Participants will be instructed to stand up from a chair, walk three meters at their usual speed, turn, walk back to the chair, and sit down. The time will be recorded.
4-meter gait speed | In the pilot part, this outcome will be assessed at baseline and within one week post-intervention. In the full RCT part, an additional measurement will be conducted within one week after the completion of the two-month follow-up period.
  This outcome will be measured in the pilot part and in the full RCT part. Participants will be required to walk 4-m distance at their usual speed twice and the faster time will be recorded.
Age | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be collected by self-reported method.
Gender | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into male and female.
Education level | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into primary school and below, middle school, high school, and bachelor's degree and above.
Marital status | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into married, single, divorced, and widowed.
Employment status | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized as employment and unemployment.
Income | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into less than 5,000, 5,000-10,000, and more than 10,000.
Living conditions | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into living alone and living with others.
Drinking status | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into never, former drinker, and current drinker.
Smoking status | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into never, former smoker, and current smoker.
Sleep duration at night | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be recorded as the hours of sleep at night.
Sleep quality | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into very poor, poor, fair, good, and very good.
Exercise habit | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into with exercise habit and without exercise habit. Exercise habit is defined as exercising at least three times per week, with each session lasting no less than 30 minutes.
Polypharmacy | This outcome will be collected at baseline.
  This outcome will be measured in the pilot part and in the full RCT part, which will be categorized into yes and no. Polypharmacy is defined as the use of five or more medications.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Xi, PhD, Principal Investigator — The University of Hong Kong
Locations (3):
- China (3):
  - Gusu District Feng Men Street Community Health Service Center, Suzhou, Jiangsu
  - Gusu District Jinchang Street Bailian Community Health Service Center, Suzhou, Jiangsu
  - Gusu District Shuang Ta Street Jinfan Community Health Service Center, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No